CLINICAL TRIAL: NCT03472352
Title: A Combination Study to Evaluate the Safety and Efficacy of an Anti-cancer Medication (A01) With Immune Cells (IC01) in Subjects With Advanced Solid Tumors
Brief Title: Safety and Efficacy of an Anticancer Medication Combined With Immune Cells in Subjects With Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hangzhou Converd Co., Ltd. (Industry)
Collaborators: The Second People's Hospital of Yibin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVD20180401
Record Dates: First submitted 2018-03-07; First posted 2018-03-21 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): The subjects will be given an anticancer medication (A01) and immune cells (IC01).
  Interventions: Biological: An anticancer medication (A01) and immune cells (IC01)

INTERVENTIONS:
Biological: An anticancer medication (A01) and immune cells (IC01) — The administration of A01 and IC01 will be performed in the Second People's Hospital of Yibin, Sichuan, China. The subjects will be observed for any side effects during this time and all the adverse events will be recorded.

SUMMARY:
This is an open-label study to evaluate the safety and efficacy of an anticancer medication (A01) with immune cells (IC01) in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion criteria:

1. Signed informed consent form must be obtained prior to any research procedures;
2. Age: 18 Years to 70 Years;
3. The patient's biological parent or child whose age ≥18 years voluntarily donates peripheral blood (100-200 ml) for the treatment, and who signs the informed consent form independently;
4. Histologically confirmed diagnosis of solid tumors;
5. Patients who have received at least one standard treatment (surgery, chemotherapy, radiotherapy, or targeted therapy) or refuse to receive standard treatments;
6. KPS > 60 points;
7. expected survival > 6 months;
8. Adequate organ function defined as: ANC≥1.0×10^9/L, PLT≥50×10^9/L, ALB≥25g/L;
9. If a subject is a female of childbearing potential, she must have a negative urine pregnancy test result.

Exclusion Criteria:

1. Patients who received chemotherapy, large-field radiotherapy or participated in other studies of anti-tumor therapy within 2 weeks before enrollment;
2. Patients who have not recovered from adverse reactions related to above-mentioned procedures;
3. Patients with two types of primary solid tumors;
4. Patients with brain metastases or bone metastases;
5. Patients with poorly controlled hypertension (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 90 mmHg), or cardiovascular and cerebrovascular diseases with clinical significance, such as cerebrovascular accident (within 6 months before signing informed consent), myocardial infarction (within 6 months before signing informed consent), unstable angina, congestive heart failure (New York Heart Association ClassⅡ or above), or severe arrhythmia which can't be controlled with drugs or have potential impact on the treatment;
6. Patients with other serious organic diseases or mental disorders;
7. Patients with systemic or active infection;
8. Patients with positive HIV test result;
9. Patients who have received an organ transplant;
10. Patients who are breastfeeding or pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
The adverse events associated with infusion of the anticancer medication or the immune cells will be assessed. | Day 0 to 4 months after the end of the study
  Incidence and duration of all the adverse events will be recorded. The severity of adverse events will be evaluated according to NCI-CTCAE v4.03 criteria.

SECONDARY OUTCOMES:
Tumor Response of the treatment in patients with advanced solid tumors. | Before treatment and Day 28 to 4 months after the end of the treatment
  Response Evaluation Criteria in Solid Tumors (RECIST) from the NCI will be used for assessment of radiographic response.